CLINICAL TRIAL: NCT07338292
Title: VIrtual Reality Induced Pain and anxiEty Relief in Outpatient UROlogical Procedures: a Post-marketing Clinical Investigation of REALICA
Brief Title: VIrtual Reality Induced Pain and anxiEty Relief in Outpatient UROlogical Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOV-UD-01-2025-VIPER_URO
Record Dates: First submitted 2025-12-23; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Urologic Diseases; Prostate Biopsy; Flexible Cystoscopy; Circumcision; Stress; Anxiety; Pain
Keywords: virtual reality; medical device
MeSH Terms: conditions — Urologic Diseases; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: REALICA® is a virtual reality viewer, designed to reduce stress and anxiety in patients during intervention and invasive procedure. This medical device effectively distracts the patient through interactive audiovisual content and promotes relaxation through guided visual and sound stimuli. The system provides in each setting for interactions designed to engage the patient's attention, consisting of simple games or activities, which require the participation of the patient through the use of the external controllers provided, who is then required to interact. The system operates anonymously, with no need to identify the patient or collect any sensitive data about the user. The device is configured as a "stand-alone" device, i.e., autonomous and without the need for wired connections to PCs or other external devices.
Who Masked: Participant
Masking Description: Control group will be treated according to clinical practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): REALICA® is a virtual reality viewer, designed to reduce stress and anxiety in patients during intervention and invasive procedure. This medical device effectively distracts the patient through interactive audiovisual content and promotes relaxation through guided visual and sound stimuli. The system provides in each setting for interactions designed to engage the patient's attention, consisting of simple games or activities, which require the participation of the patient through the use of the external controllers provided, who is then required to interact. The system operates anonymously, with no need to identify the patient or collect any sensitive data about the user. The device is configured as a "stand-alone" device, i.e., autonomous and without the need for wired connections to PCs or other external devices.
  Interventions: Device: REALICA
- Control group (Active Comparator): Control group will be treated according to clinical practice.
  Interventions: Other: Clinical Practice

INTERVENTIONS:
Device: REALICA — REALICA® is a virtual reality viewer, designed to reduce stress and anxiety in patients during intervention and invasive procedure. This medical device effectively distracts the patient through interactive audiovisual content and promotes relaxation through guided visual and sound stimuli. The system provides in each setting for interactions designed to engage the patient's attention, consisting of simple games or activities, which require the participation of the patient through the use of the external controllers provided, who is then required to interact. The system operates anonymously, with no need to identify the patient or collect any sensitive data about the user. The device is configured as a "stand-alone" device, i.e., autonomous and without the need for wired connections to PCs or other external devices.
  Arms: Virtual reality
Other: Clinical Practice — Patients in the Control group will receive topical anesthesia, without application of virtual viewer.
  Arms: Control group

SUMMARY:
Though the efficacy of VRH is documented in various outpatient urological procedures and has provided promising preliminary information in prostate biopsy, its systematic use in urology remains poorly studied. Considering the potential of invasive urological procedures to induce significant patient discomfort, the application of innovative immersive approaches, such as those offered by medical devices, could lead to an overall clinical benefit. Among these, REALICA® (available from https://REALICA.io/en/), a class I CE medical device, widely used in hospitals and validated by numerous studies, represents a valuable resource in urology, supported by high satisfaction rates received in abdominal surgery and extracorporeal lithotripsy

DETAILED DESCRIPTION:
Routine outpatient urological procedures, including circumcision, prostate biopsy, and flexible cystoscopy, despite being minimally invasive, are often accompanied by high levels of preoperative anxiety and anticipatory pain. Inadequate management of such symptoms not only compromises patient experience and compliance with future treatments, but can also lead to procedural stress-related complications such as intraoperative hypertension and tachycardia. Consequently, the identification and implementation of effective strategies to mitigate these events are of primary importance. Traditionally, pharmacological sedatives are used to alleviate anxiety and pain; however, these can cause adverse events, require intensive monitoring, and increase healthcare costs, slowing patient turnover in outpatient settings. For this reason, non-pharmacological strategies, known as "digital sedation" and including virtual reality, music therapy, and biofeedback, are emerging as effective options to optimize patient comfort while limiting exposure to sedative drugs. In particular, medical hypnosis promotes a state of deep relaxation and focused attention, demonstrating its applicability in the management of chronic and procedural pain, as well as in anxiety reduction in various clinical settings. Among these strategies, Virtual Reality Hypnosis (VRH) combines interactive immersion in three-dimensional environments with guided hypnotic scripts, leveraging distraction and suggestion mechanisms to modulate the perception of anxiety and pain. Recent systematic reviews and meta-analyses have corroborated the effectiveness of VRH in heterogeneous contexts (bronchoscopy, interventional radiology, dentistry, and orthopedics) with significant reductions in subjective pain scores and autonomic stress parameters (heart rate, blood pressure). For example, Ahmad et al. (2020) found an average 20-30% improvement in pain and anxiety levels in cancer patients undergoing invasive procedures [8], while Georgescu et al. (2020) documented an effect size up to 0.8 for VRH analgesia in procedural settings. Zheng et al. (2022) further demonstrated an increase of over 15% in nociceptive pain threshold and favorable modulation of autonomic functions in healthy volunteers. Finally, Teh, Jia J et al. (2024), including 23 randomized trials, highlighted an average 25% decrease in intra-procedural pain and significant comfort improvement, reinforcing VRH's potential as a digital sedation tool. In the urological field, controlled studies have utilized VRH sets during flexible cystoscopy, achieving significant reductions in anxiety, pain, and hemodynamic parameters compared to controls; analogous results have been confirmed by technical feasibility and symptom decrease in rigid cystoscopies. The integration of VRH masks in minimally invasive functional urological interventions has achieved satisfaction rates exceeding 90% and reductions of up to 35% in self-reported pain. Further preliminary studies on transperineal prostate biopsy have also shown trends towards a decrease in anxiety state and increased willingness to repeat the procedure, while an ongoing trial is evaluating the effectiveness of VRH headphones on anxiety and comfort during transrectal biopsy. Finally, a recent mini-review highlighted the potential of VRH as a supportive tool for local anesthesia in outpatient urological procedures, as well as the need for further randomized studies to define specific protocols.

ELIGIBILITY:
Inclusion Criteria:

* Male/female with age ≥ 18 years
* Patient who are undergoing one of the interventions mentioned in the study for the first time;
* Eligibility for minimally invasive ambulatory urological procedures, possibly requiring vascular access (circumcision, prostate biopsy, flexible cystoscopy);
* Ability to understand instructions and complete study questionnaires;
* Signed informed consent.

Exclusion Criteria:

* Absolute contraindications to the planned urological procedure (e.g., active urinary tract infection, anatomical urethral abnormalities);
* Recent urological manipulations (e.g., urethral dilation, bladder biopsy, insertion or removal of a double-J stent);
* Medical contraindications to the use of virtual reality, including uncontrolled photosensitive epilepsy and relevant neurological, ophthalmologic, or otolaryngologic disorders;
* Presence of severe psychiatric disorders or major cardiovascular diseases that may interfere with study participation;
* Previous adverse reactions to virtual reality exposure;
* Use of analgesic medications within 24 hours prior to the procedure;
* Use of drugs that may alter consciousness or impair the ability to complete psychological assessments;
* Severe communication disabilities or significant hearing impairment that would prevent completion of questionnaires.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety reduction | Through study completion, an average of 1 year
  Evaluate the impact of immersive virtual reality on reducing anxiety, in patients undergoing minimally invasive ambulatory urological procedures, such as prostate biopsy, flexible cystoscopy, and circumcision using validated patient-reported scales STAI (State-Trait Anxiety Inventory), before and after invasive procedure.
  The minimum value is 1 = almost never and the maximum value is 4=almost always

SECONDARY OUTCOMES:
Intensity of pain | Through study completion, an average of 1 year
  Assess the intensity of pain perceived by patients during the procedure with the use of REALICA. Measurement of pain intensity perceived by patients during the procedure (T1) with the use of a virtual reality headset, assessed through validated scale as the Visual Analog Scale (VAS). The minimum value is Left = no pain; the maximum value is right = the worst pain imaginable
Intensity of pain | Through study completion, an average of 1 year
  Assess the intensity of pain perceived by patients during the procedure with the use of REALICA. Measurement of pain intensity perceived by patients during the procedure (T1) with the use of a virtual reality headset, assessed through validated scale as the Numeric Rating Scale (NRS).
  The minimum value is 0 = no pain, the maximum value is 10 = the worst pain imaginable.
Pain levels | Through study completion, an average of 1 year
  Evaluation of the reduction in pain levels associated with minimally invasive ambulatory urological procedures attributable to the use of virtual reality, using validated patient-reported scale VAS (Visual Analog Scale). The minimum value is Left = no pain; the maximum value is right = the worst pain imaginable
Pain levels | Through study completion, an average of 1 year
  Evaluation of the reduction in pain levels associated with minimally invasive ambulatory urological procedures attributable to the use of virtual reality, using validated patient-reported scale NRS (Numeric Rating Scale). The minimum value is 0 = no pain, the maximum value is 10 = the worst pain imaginable.
Feasibility and acceptability of REALICA® | Through study completion, an average of 1 year
  Evaluation of feasibility and acceptability of virtual reality headset use in the intervention group, based on the proportion of patients who tolerate and complete the VR intervention, along with feedback collected from patients and healthcare professionals via the modified System Usability Scale (SUS) questionnaires and Likert scales, which will be administered to patients and staff upon completion of the procedure. The minimum value is 1 = Strongly agree, the maximum value is 5 = strongly disagree.
Patient Satisfaction Questionnaire | Through study completion, an average of 1 year
  Assess patient satisfaction with the virtual reality intervention using the Patient Satisfaction Questionnaire (PSQ). The minimum value is 1 = Strongly agree, the maximum value is 5 = strongly disagree.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto IRCCS, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Deniz Dogan S, Yurtseven S, Arslan S. The Effect of Preoperative Pain, Fear, and Anxiety on Postoperative Pain in Urological Surgery Patients: A Descriptive and Correlational Study. J Perianesth Nurs. 2024 Apr;39(2):202-206. doi: 10.1016/j.jopan.2023.07.013. Epub 2023 Nov 3. PMID 37921714
- [Result] Jiao D. Advancing personalized digital therapeutics: integrating music therapy, brainwave entrainment methods, and AI-driven biofeedback. Front Digit Health. 2025 Feb 25;7:1552396. doi: 10.3389/fdgth.2025.1552396. eCollection 2025. PMID 40070544
- [Result] Terzulli C, Chauvin C, Champagnol Di-Liberti C, Faisan S, Goffin L, Gianesini C, Graff D, Dufour A, Laroche E, Salvat E, Poisbeau P. Virtual reality hypnosis diminishes experimental cold pain and alters autonomic responses. Front Pain Res (Lausanne). 2023 Nov 2;4:1237090. doi: 10.3389/fpain.2023.1237090. eCollection 2023. PMID 38028428
- [Result] Rizzo MG Jr, Costello JP 2nd, Luxenburg D, Cohen JL, Alberti N, Kaplan LD. Augmented Reality for Perioperative Anxiety in Patients Undergoing Surgery: A Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2329310. doi: 10.1001/jamanetworkopen.2023.29310. PMID 37589975
- [Result] Ahmad M, Bani Mohammad E, Anshasi HA. Virtual Reality Technology for Pain and Anxiety Management among Patients with Cancer: A Systematic Review. Pain Manag Nurs. 2020 Dec;21(6):601-607. doi: 10.1016/j.pmn.2020.04.002. Epub 2020 May 15. PMID 32423641
- [Result] Georgescu R, Fodor LA, Dobrean A, Cristea IA. Psychological interventions using virtual reality for pain associated with medical procedures: a systematic review and meta-analysis. Psychol Med. 2020 Aug;50(11):1795-1807. doi: 10.1017/S0033291719001855. Epub 2019 Aug 28. PMID 31456530
- [Result] Terzulli C, Melchior M, Goffin L, Faisan S, Gianesini C, Graff D, Dufour A, Laroche E, Chauvin C, Poisbeau P. Effect of Virtual Reality Hypnosis on Pain Threshold and Neurophysiological and Autonomic Biomarkers in Healthy Volunteers: Prospective Randomized Crossover Study. J Med Internet Res. 2022 Jul 29;24(7):e33255. doi: 10.2196/33255. PMID 35904872
- [Result] Teh JJ, Pascoe DJ, Hafeji S, Parchure R, Koczoski A, Rimmer MP, Khan KS, Al Wattar BH. Efficacy of virtual reality for pain relief in medical procedures: a systematic review and meta-analysis. BMC Med. 2024 Feb 14;22(1):64. doi: 10.1186/s12916-024-03266-6. PMID 38355563
- [Result] Ketsuwan C, Matang W, Ratanapornsompong W, Sangkum P, Phengsalae Y, Kongchareonsombat W, Jongwannasiri M. Prospective randomized controlled trial to evaluate effectiveness of virtual reality to decrease anxiety in office-based flexible cystoscopy patients. World J Urol. 2022 Oct;40(10):2575-2581. doi: 10.1007/s00345-022-04142-9. Epub 2022 Sep 1. PMID 36048232
- [Result] Luczak M, Nowak L, Chorbinska J, Galik K, Kielb P, Laszkiewicz J, Tukiendorf A, Koscielska-Kasprzak K, Malkiewicz B, Zdrojowy R, Szydelko T, Krajewski W. Influence of Virtual Reality Devices on Pain and Anxiety in Patients Undergoing Cystoscopy Performed under Local Anaesthesia. J Pers Med. 2021 Nov 16;11(11):1214. doi: 10.3390/jpm11111214. PMID 34834565
- [Result] Geretto P, De Cillis S, Candela L, Germain T, Vienney N, Felber M, Phe V. Integrating a Virtual Reality Mask in Functional Urological Surgeries Under Local Anesthesia: A Prospective Cohort Study on Utility and Satisfaction. Urology. 2025 Feb;196:93-99. doi: 10.1016/j.urology.2024.11.007. Epub 2024 Nov 14. PMID 39547279
- [Result] Perucchini F, Baumeister P, Fankhauser CD. Beyond Anesthesia: A Mini Review of Virtual Reality as an Adjunct in Urological Procedures. Eur Urol Focus. 2025 May;11(3):511-514. doi: 10.1016/j.euf.2025.01.007. Epub 2025 Jan 22. PMID 39848858
- [Result] Candela L, Ventimiglia E, Corrales M, Sierra Del Rio A, Villa L, Goumas IK, Salonia A, Montorsi F, Doizi S, Traxer O. The Use of a Virtual Reality Device (HypnoVR) During Extracorporeal Shockwave Lithotripsy for Treatment of Urinary Stones: Initial Results of a Clinical Protocol. Urology. 2023 May;175:13-17. doi: 10.1016/j.urology.2023.01.048. Epub 2023 Feb 15. PMID 36796544
- [Result] Carannante F, Capolupo GT, Miacci V, Ferri C, Agro FE, Caricato M, D'Agostino F. The effect of virtual reality hypnosis (HypnoVR) in patients undergoing inguinal hernia repair under local anesthesia. A preliminary report. Langenbecks Arch Surg. 2024 Oct 29;409(1):329. doi: 10.1007/s00423-024-03524-4. PMID 39470831
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/37921714/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40070544/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38028428/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37589975/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32423641/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31456530/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35904872/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38355563/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36048232/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34834565/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39547279/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39848858/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39470831/